CLINICAL TRIAL: NCT05844215
Title: Role of MMP-9, TIMP-1 as Markers of Lung Imaging and Functional Abnormality of COVID-19
Brief Title: MMP-9, TIMP-9 in Lung Imaging and Functional of COVID-19
Status: Completed | Type: Observational
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Alfian Nur Rosyid, Doctoral Student, Faculty of Medicine, Universitas Airlangga
Other Study IDs: 206/RSUA
Record Dates: First submitted 2023-04-29; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Infection; COVID-19; Extracellular Matrix Alteration
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — A blood sample was taken from the sample study during admission (after the patient agreed to join the study and signed the informed consent). Blood is stored in a refrigerator at -80 degrees Celsius. After all study samples have been collected, the blood is removed from the refrigerator and examined by ELISA. The distance between the first and last blood samples was about six months, and then a sample examination was carried out simultaneously. MMP-9 and TIMP-1 were checked using ELISA from sample blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Severe: Non-severe groups consisted of mild and moderate severity of COVID-19. Mild-degree are patients with symptoms of COVID-19 but do not require oxygen with normal X-ray images. Moderate-degree are patients with symptoms of COVID-19 that require a low oxygen flow rate with minimal pneumonia on chest X-Ray.
  Interventions: Diagnostic Test: MMP-9 and TIMP-1
- Severe: Severe groups consisted of Severe and Critical Ill of COVID-19. Severe-degree are patients that require high oxygen flow rate with diffuse lung infiltrates. Critical-Ill are COVID-19 patients that suffered shock sepsis or respiratory failure.
  Interventions: Diagnostic Test: MMP-9 and TIMP-1

INTERVENTIONS:
Diagnostic Test: MMP-9 and TIMP-1 — Examine level of serum MMP-9 and TIMP-1

SUMMARY:
This study aims to determine the role of the extracellular matrix in lung abnormalities in COVID-19 patients. Anatomical abnormalities of the lungs can be observed by the presence of abnormalities on a chest x-ray that is scored using the Brixia index. The presence of COVID-19 pneumonia can impact oxygenation disorders. It is hoped that knowing the relationship between biomarkers that affect the extracellular matrix and anatomical and functional abnormalities can open up new insights into new therapeutic opportunities. The balance of MMP-9 and TIMP-1 has been studied in relation to several lung diseases other than COVID-19.

DETAILED DESCRIPTION:
Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV2), which has different degrees of severity, is the cause of Coronavirus Disease 2019 (COVID-19). Over 97% of COVID-19 patients make a full recovery. Inflammation increases when COVID-19 severity increases. The lungs and endothelium will suffer harm when different pro-inflammatory cytokines are released. A cytokine storm is started when many immune cells produce cytokines and chemokines. The pro-inflammatory cytokine can increase angiogenesis, vascular permeability, keratin proliferation, and collagen production. Lung lesions are affected by certain disorders. In COVID-19 patients, angiogenesis, fibroblast activation, and collagen deposition all contribute to the repair of the lungs. The pathological outcome of acute or chronic interstitial pulmonary disease is lung fibrosis, characterized by abnormal collagen and extracellular matrix (ECM) deposition, the persistence of fibroblasts, failure of alveolar re-epithelization, and destruction of normal pulmonary architecture. The breakdown or buildup of ECM is influenced by the ratio of matrix metalloproteinase (MMP) and tissue inhibitor matrix metalloproteinase (TIMP). TIMP distribution, not MMP distribution, was the primary contributor to lung fibrosis. MMP expression is increased by the production of several hormones, cytokines (IL-1, IL-6), growth factors (TGF, TNF-), platelet-derived growth factor (PDGF), and basic fibroblast growth factor (bFGF).

ECM assistance is required for the alveoli to function normally. Excessive ECM breakdown and aberrant ECM remodelling are the root causes of many respiratory conditions, including pulmonary fibrosis. ECM buildup destroys the alveolar process, particularly by impairing alveolar-capillary diffusion. On radiological images, lung abnormalities can be seen as pneumonia in the bilateral ground-glass opacity basal, which results in hypoxia. In the lower portion, bilateral abnormalities predominated. COVID-19 ARDS, hypoxemia, bilateral infiltrates, and reduced lung compliance were the hallmarks of pneumonia type H. Despite the limited sensitivity, plain chest X-rays can detect lung abnormalities in COVID-19; they are inexpensive and simple. New infiltrates on chest radiographs were used to make the diagnosis of pneumonia.

Biomarkers of pulmonary interstitial abnormalities have received limited attention in the literature, including investigations on MMP and TIMP for lung abnormalities in COVID-19 patients. One of the MMP gelatinase family's more complicated forms, MMP-9, can break down ECM components. MMP-9 increases collagen and cytokine production, fibroblast migration, and TGF- stimulation. MMP-9 is among the MMPs that TIMP1 effectively inhibits. TIMP-1 binds to pro- or latent MMP-9. For ECM proteolysis to occur, MMP and TIMP must coexist in equilibrium. This study aimed to ascertain how MMP-9 and TIMP-1 affected abnormal chest X-rays, poor oxygenation, severity, and death.

Blood is taken from hospitalized COVID-19 patients to measure the serum concentrations of MMP-9 and TIMP-1. At the time of hospital admission, three reviewers assessed the severity after chest X-Rays, followed by a BRIXIA score. At the time of hospital discharge, patients were evaluated. The levels of MMP-9 and TIMP-1 were compared to Brixia scores, oxygen consumption, severity, and death.

ELIGIBILITY:
Inclusion Criteria:

* The patient is infected with COVID-19 with positive RT-PCR Swab results
* Age 21-70 years
* Men or Women
* Various degrees of severity (mild, moderate, severe, critical) and comorbidities
* the Chest X-ray was done
* Willing to participate in research (signing informed consent)

Exclusion Criteria:

* The patient is TB active or has been treated for pulmonary TB
* Patients with a history of ILD clinically
* Patients with a history of asthma or COPD
* Pregnant women
* HIV/AIDS patients

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized COVID-19 patients in Universitas Airlangga Surabaya, Indonesia, proven by positive swab RT-PCR COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Anatomical abnormalities of the lungs. | Chest X-Ray checked 2-4 hours during admission in emergency room.
  Anatomical of the lung measured by Chest X-ray abnormality, scored by Brixia Index.
Functional abnormalities of the lungs. | Oxygen use and blood gas analysis checked 1-2 hours during admission in emergency room.
  Functional of the lung measured by the oxygen used and Blood Gas Analysis.

SECONDARY OUTCOMES:
Severity | Severity measured when patient hospitalized at first time during inclusion of study (4-6 hours after admission).
  Severity is the degree of severity at the time of admission to the hospital.
Mortality | Mortality measured when patient out from hospital during the study (end of study).
  Mortality is measured by the condition of being discharged from the hospital, whether dead or alive.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Amin, Prof., Principal Investigator — Airlangga University Faculty of Medicine: Universitas Airlangga Fakultas Kedokteran
Locations (1):
- Universitas Airlangga Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Researchers have not yet decided to share data, but they do not rule out other researchers wishing to be able to access primary research data. Other researchers can contact the principal investigator via email.

REFERENCES:
- [Background] Lingeswaran M, Goyal T, Ghosh R, Suri S, Mitra P, Misra S, Sharma P. Inflammation, Immunity and Immunogenetics in COVID-19: A Narrative Review. Indian J Clin Biochem. 2020 Jul;35(3):260-273. doi: 10.1007/s12291-020-00897-3. Epub 2020 Jun 6. PMID 32641873
- [Background] Ojo AS, Balogun SA, Williams OT, Ojo OS. Pulmonary Fibrosis in COVID-19 Survivors: Predictive Factors and Risk Reduction Strategies. Pulm Med. 2020 Aug 10;2020:6175964. doi: 10.1155/2020/6175964. eCollection 2020. PMID 32850151
- [Background] Gill SE, Parks WC. Metalloproteinases and their inhibitors: regulators of wound healing. Int J Biochem Cell Biol. 2008;40(6-7):1334-47. doi: 10.1016/j.biocel.2007.10.024. Epub 2007 Oct 26. PMID 18083622
- [Background] Signoroni A, Savardi M, Benini S, Adami N, Leonardi R, Gibellini P, Vaccher F, Ravanelli M, Borghesi A, Maroldi R, Farina D. BS-Net: Learning COVID-19 pneumonia severity on a large chest X-ray dataset. Med Image Anal. 2021 Jul;71:102046. doi: 10.1016/j.media.2021.102046. Epub 2021 Mar 31. PMID 33862337
- [Background] Gu Y, Wang D, Chen C, Lu W, Liu H, Lv T, Song Y, Zhang F. PaO2/FiO2 and IL-6 are risk factors of mortality for intensive care COVID-19 patients. Sci Rep. 2021 Apr 1;11(1):7334. doi: 10.1038/s41598-021-86676-3. PMID 33795768
- [Background] Elkington PT, Friedland JS. Matrix metalloproteinases in destructive pulmonary pathology. Thorax. 2006 Mar;61(3):259-66. doi: 10.1136/thx.2005.051979. Epub 2005 Oct 14. PMID 16227332
- [Background] D Avila-Mesquita C, Couto AES, Campos LCB, Vasconcelos TF, Michelon-Barbosa J, Corsi CAC, Mestriner F, Petroski-Moraes BC, Garbellini-Diab MJ, Couto DMS, Jordani MC, Ferro D, Sbragia L, Joviliano EE, Evora PR, Carvalho Santana R, Martins-Filho OA, Polonis K, Menegueti MG, Ribeiro MS, Auxiliadora-Martins M, Becari C. MMP-2 and MMP-9 levels in plasma are altered and associated with mortality in COVID-19 patients. Biomed Pharmacother. 2021 Oct;142:112067. doi: 10.1016/j.biopha.2021.112067. Epub 2021 Aug 20. PMID 34449310
- [Background] Guizani I, Fourti N, Zidi W, Feki M, Allal-Elasmi M. SARS-CoV-2 and pathological matrix remodeling mediators. Inflamm Res. 2021 Aug;70(8):847-858. doi: 10.1007/s00011-021-01487-6. Epub 2021 Jul 20. PMID 34286362